CLINICAL TRIAL: NCT01435109
Title: Patient and Provider Interventions for Managing Osteoarthritis in Primary Care
Acronym: PRIMO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Health Services Research
Other Study IDs: Pro00022836; R01AR059673 (NIH)
Record Dates: First submitted 2011-09-07; First posted 2011-09-15 (Estimated); Last update posted 2016-06-08 (Estimated); Status verified 2016-06

CONDITIONS: Osteoarthritis
Keywords: Osteoarthritis; Exercise; Diet; Coping Skills; Education, Medical
MeSH Terms: conditions — Osteoarthritis; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Usual Care (No Intervention)
- Patient Behavioral Intervention (Experimental): Patients receive a 12-month intervention consisting of monthly phone calls focusing on exercise, weight management, and cognitive behavioral pain management.
  Interventions: Behavioral: Patient Behavioral Intervention for OA
- Provider Intervention (Experimental): Primary care providers receive patient-specific osteoarthritis information and treatment recommendations at the point of clinical care.
  Interventions: Behavioral: Provider Intervention for OA
- Patient and Provider Interventions (Experimental): Patients receive a 12-month intervention consisting of monthly phone calls focusing on exercise, weight management, and cognitive behavioral pain management; primary care providers receive patient-specific osteoarthritis information and treatment recommendations at the point of clinical care.
  Interventions: Behavioral: Combined Patient and Provider Interventions for OA

INTERVENTIONS:
Behavioral: Patient Behavioral Intervention for OA — Patients receive a 12-month intervention consisting of monthly phone calls focusing on exercise, weight management, and cognitive behavioral pain management.
  Arms: Patient Behavioral Intervention
Behavioral: Provider Intervention for OA — Primary care providers receive patient-specific osteoarthritis information and treatment recommendations at the point of clinical care.
  Arms: Provider Intervention
Behavioral: Combined Patient and Provider Interventions for OA — Patients receive a 12-month intervention consisting of monthly phone calls focusing on exercise, weight management, and cognitive behavioral pain management; primary care providers receive patient-specific osteoarthritis information and treatment recommendations at the point of clinical care.
  Arms: Patient and Provider Interventions

SUMMARY:
Osteoarthritis (OA) is one of the most common chronic conditions and a leading cause of pain and disability among adults. Many adults with OA have significant pain and functional limitations, even though they receive some medical care for their OA. Efforts are needed to help adults improve OA-related outcomes. This study will examine three different approaches for helping adults manage their OA-related symptoms. The study will compare a patient-based intervention (involving exercise, weight management, and cognitive behavioral pain management), a provider-based intervention (involving provision of patient-specific recommendations for care, based on evidence-based guidelines), and a combination of the two interventions, relative to usual care among patients with hip and/or knee osteoarthritis. The interventions are relatively low cost and easy to disseminate, with the patient component being telephone based. This study will provide novel, valuable information of the effectiveness (and cost-effectiveness) of these three interventions in the context of real-world clinical settings.

DETAILED DESCRIPTION:
Evidence-based guidelines emphasize that adequate management of osteoarthritis (OA) requires a combination of both medical and behavioral modalities. However, many of the recommended guidelines are not regularly incorporated into clinical practice, and the recommended behavioral strategies (e.g. exercise and weight management) are not practiced by most patients. Prior studies have examined strategies for improving patient behaviors to manage OA-related symptoms, but few studies have examined provider-based interventions specifically for patients with OA, or combinations of patient- and provider-based interventions. The objective of this study is to compare a patient-based intervention (involving exercise, weight management, and cognitive behavioral pain management), a provider-based intervention (involving provision of patient-specific recommendations for care, based on evidence-based guidelines), and a combination of the two interventions, relative to usual care. This study will provide novel, valuable information of the effectiveness (and cost-effectiveness) of these three interventions in the context of real-world clinical settings.

This will be a randomized controlled trial involving the following four study arms: 1) Patient Behavioral Intervention for OA Only, 2) Provider Intervention for OA Only, 3) Patient Behavioral Intervention + Provider Intervention for OA, and 4) Usual Care Control (no intervention). Approximately 10 primary care practices in the Duke Primary Care Research Consortium (PCRC) will be randomized to either the Provider Intervention or Provider Control group. Within each clinic, patients with symptomatic knee and/or hip OA (n=560 total) will be randomly assigned to either the Patient Intervention or Patient Control group. Participants will be equally allocated between the four study groups, with randomization stratified according to gender and race (white/non-white).

The patient behavioral intervention will be a twelve-month program that includes the following elements: written educational materials (focused on exercise, weight management, and cognitive behavioral pain management), an exercise video tailored for patients with lower extremity OA, and telephone calls by a counselor to support behavior change. All participants in the study will continue with any other usual medical care they receive for OA. The provider intervention will involve giving information on patients' OA symptoms and treatment, as well as patient-specific evidence-based recommendations for care. Providers will have access to this information, as well as facilitated referrals for patient-specific treatment recommendations (e.g. physical therapy, orthopedics), at the point of clinical care.

The primary time point for outcome assessment will be at 12-months. The investigators will also assess a limited set of outcomes via telephone at 6-months, 18-months, and 24-months. Following completion of study follow-up assessments, participants who were not assigned to one of the two Participant arms will be given the materials for that intervention, and health care providers who were not part of one of the two Provider arms will be given the information involved in that intervention. The primary outcome will be the Western Ontario and McMasters Universities Osteoarthritis Index (WOMAC). Secondary outcomes will include objective physical function (Short Physical Performance Test) and depressive symptoms (PHQ-8). The main study analyses will compare outcomes between the four study groups. The investigators will also assess the cost-effectiveness of the interventions.

ELIGIBILITY:
Inclusion Criteria:

* Radiographic evidence of hip OA and/or radiographic evidence of or meets clinical criteria for knee OA
* Current joint (hip and/or knee) symptoms
* BMI >= 25
* Physically inactive

Exclusion Criteria:

* Diagnosis of rheumatoid arthritis, fibromyalgia, or other systemic rheumatic disease
* Diagnosis of a motor neuron disease, Parkinson's disease, multiple sclerosis, or Paget's disease
* Diagnosis of metastatic cancer
* Hospitalized for a stroke, myocardial infarction or coronary artery revascularization in the past 3 months
* On waiting list for or planning arthroplasty
* Total joint replacement (hip or knee) surgery, other hip or knee surgery, meniscus tear (verified by MRI), or ACL tear in the past 6 months
* History of gout in hip or knee
* Quadriplegia or paraplegia
* Active diagnosis of psychosis or serious personality disorder
* Diagnosis of dementia or other memory loss condition
* Current, uncontrolled substance abuse disorder
* Severly impaired speech or hearing (patients must be able to respond to phone calls)
* No access to a telephone
* Inability to understand and speak English
* Blindness
* Resident in nursing home
* Serious / terminal illness as indicated by referral to hospice or palliative care
* For females: currently pregnant or planning to become pregnant
* No visit to their Duke primary health care provider in the last 18 months
* Participating in another OA intervention of other lifestyle change study
* Other self-reported medical problem that would prohibit participation in the study
* Other health condition or personal issue judged by a study team member or primary care physician to make the patient inappropriate for study participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 537 (Actual)
Dates: Start 2011-07; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Change in the Western Ontario and McMasters Universities Osteoarthritis Index (WOMAC) from Baseline to 12-months. | Baseline and 12-months
Change in the Western Ontario and McMasters Universities Osteoarthritis Index (WOMAC) at 18-months post Baseline. | post Baseline,18-months
Change in the Western Ontario and McMasters Universities Osteoarthritis Index (WOMAC) at 24-months post Baseline. | post Baseline, 24-months

SECONDARY OUTCOMES:
Change in the Short Physical Performance Test Protocol from Baseline to 12-months. | Baseline and 12-months
Change in the Patient Health Questionnaire (PHQ-8) from Baseline to 12-months. | Baseline and 12-months

CONTACTS AND LOCATIONS:
Overall Officials: Kelli D Allen, PhD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

REFERENCES:
- [Background] Allen KD, Bosworth HB, Brock DS, Chapman JG, Chatterjee R, Coffman CJ, Datta SK, Dolor RJ, Jeffreys AS, Juntilla KA, Kruszewski J, Marbrey LE, McDuffie J, Oddone EZ, Sperber N, Sochacki MP, Stanwyck C, Strauss JL, Yancy WS Jr. Patient and provider interventions for managing osteoarthritis in primary care: protocols for two randomized controlled trials. BMC Musculoskelet Disord. 2012 Apr 24;13:60. doi: 10.1186/1471-2474-13-60. PMID 22530979
- [Background] Allen KD, Bosworth HB, Chatterjee R, Coffman CJ, Corsino L, Jeffreys AS, Oddone EZ, Stanwyck C, Yancy WS Jr, Dolor RJ. Clinic variation in recruitment metrics, patient characteristics and treatment use in a randomized clinical trial of osteoarthritis management. BMC Musculoskelet Disord. 2014 Dec 6;15:413. doi: 10.1186/1471-2474-15-413. PMID 25481809
- [Derived] Allen KD, Oddone EZ, Coffman CJ, Jeffreys AS, Bosworth HB, Chatterjee R, McDuffie J, Strauss JL, Yancy WS Jr, Datta SK, Corsino L, Dolor RJ. Patient, Provider, and Combined Interventions for Managing Osteoarthritis in Primary Care: A Cluster Randomized Trial. Ann Intern Med. 2017 Mar 21;166(6):401-411. doi: 10.7326/M16-1245. Epub 2017 Jan 17. PMID 28114648